CLINICAL TRIAL: NCT00384150
Title: A Phase III, Open-Label, Multicenter, Single-Arm, Retreatment Study of Galiximab in Combination With Rituximab for Subjects With Relapsed, Follicular Non-Hodgkin's Lymphoma Who Previously Responded on Study 114-NH-301
Brief Title: Retreatment Study of Galiximab + Rituximab in Follicular Non-Hodgkin's Lymphoma (NHL)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment challenges due to changes in standards of care resulted in premature termination. No safety or efficacy events factored into this action.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114-NH-302
Record Dates: First submitted 2006-10-04; First posted 2006-10-05 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-10

CONDITIONS: Lymphoma, Non-Hodgkin's
Keywords: galiximab; antibody; refractory; follicular; relapsed; NHL; rituximab; retreatment
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — galiximab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: galiximab in combination with rituximab — galiximab (500 mg/m2 IV) in combination with rituximab (375 mg/m2 IV)once weekly for 4 weeks.

SUMMARY:
This is a Phase III, multicenter, global, open-label, single-arm, retreatment study of an investigational drug called galiximab in combination with an approved drug called rituximab in subjects with relapsed or refractory, follicular NHL who demonstrated a response on Study 114-NH-301 with a time-to-progression >=6 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Demonstrated a response (CR, CRu, or PR) on Study 114-NH-301 (Galiximab in combination with Rituximab compared with Rituximab in combination with Placebo) and then relapsed or progressed with a TTP >=6 months. Relapsed disease is defined as documented disease progression using the International Workshop Response Criteria (IWRC).
* Bidimensionally measurable disease with at least 1 lesion >=2.0 cm in a single dimension.
* Acceptable hematologic, hepatic, and renal function.

Key Exclusion Criteria:

* Any lymphoma therapy between Final Visit on Study 114-NH-301 and Study Day 1 of this retreatment study.
* Chronic or intermittent corticosteroids for inflammatory or autoimmune disorders within 3 weeks prior to Study Day 1.
* Transfusion-dependent subjects.
* Presence of central nervous system (CNS) lymphoma.
* Histologic transformation.
* Presence of pleural or peritoneal effusion with positive cytology for lymphoma.
* Another primary malignancy requiring active treatment.
* Serious nonmalignant disease (e.g., congestive heart failure, hydronephrosis); active uncontrolled bacterial, viral, or fungal infections; or other conditions that would compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
* New York Heart Association Class III or IV cardiac disease or myocardial infarction within 6 months prior to Study Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety measures include: adverse event rates, clinical laboratory results, development of anti-galiximab and human anti-chimeric antibodies | Study period is approx. 2 years

SECONDARY OUTCOMES:
Pharmacokinetics | Study period is approx. 2 years
To further characterize the efficacy profile of galiximab in combination with rituximab | Study period is approx. 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen